CLINICAL TRIAL: NCT02228993
Title: Quality of Recovery Following Awake Craniotomy Versus Craniotomy Performed Under General Anesthesia
Brief Title: Quality of Recovery Awake Versus Asleep Craniotomy
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, John Bebawy, Associate Professor of Anesthesiology & Neurological Surgery, Northwestern University
Other Study IDs: STU00096969
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Awake Craniotomy
- General Anesthesia Craniotomy

SUMMARY:
Awake craniotomy (AC) is an anesthetic and surgical technique commonly used to resect tumors involving or adjacent to the eloquent or motor cortices, those portions of the brain that are responsible for language and motor skills, respectively. By mapping those areas of the brain that are necessary for such functions, the neurosurgeon is able to avoid resection of cortical tissue that might compromise the patient's abilities to speak or move, hence preserving neurologic function. AC is often accomplished by direct cortical stimulation or inhibition, while maintaining the patient's ability to interact with the operative team. The anesthetic technique often involves a regional (scalp) block combined with intraoperative intravenous mild sedation. In some reported instances of AC, no cortical mapping is performed, and the technique is performed solely because it is thought that AC leads to a better recovery profile (less pain, better neurologic outcome, and shorter hospital stay) than craniotomy performed under general anesthesia.

The Quality of Recovery Score (QoR-40) is a validated, multi-parameter instrument that has been used in various postoperative populations to assess the overall satisfaction and well-being of patients having undergone anesthesia and surgery. Leslie et al. have reported that the QoR-40 is a valid tool in assessing neurosurgical patients, but a direct comparison between AC patients and general anesthesia craniotomy (GAC) patients using this tool has never been performed.

AC may also be associated with better 30 and 90 day multi-parameter outcomes than GAC. The well-validated Acute Short Form (SF-12) health survey, an abbreviated version of the SF-36, consists of 12 items. It measures two domains, including mental and physical component summaries (mental component summary and physical composite score, respectively).

Hypothesis:

Awake craniotomy for tumor resection is associated with a better multi-parameter quality of recovery in the immediate postoperative period, and better 30 and 90 day quality of life outcomes, than craniotomy performed under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult non-pregnant patients (age ≥ 18 years) undergoing AC or GAC for elective supratentorial tumor resection.

Exclusion Criteria:

* Patients under 18 years of age, non-English speaking, pregnancy, unable to obtain written informed consent, infratentorial tumors.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult non-pregnant patients (age ≥ 18 years) undergoing Awake Craniotomy or General Anesthesia Craniotomy for elective supratentorial tumor resection.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Quality of Recovery (QoR-40) score | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Wrede KH, Stieglitz LH, Fiferna A, Karst M, Gerganov VM, Samii M, von Gosseln HH, Ludemann WO. Patient acceptance of awake craniotomy. Clin Neurol Neurosurg. 2011 Dec;113(10):880-4. doi: 10.1016/j.clineuro.2011.06.010. Epub 2011 Jul 23. PMID 21782320
- [Background] Serletis D, Bernstein M. Prospective study of awake craniotomy used routinely and nonselectively for supratentorial tumors. J Neurosurg. 2007 Jul;107(1):1-6. doi: 10.3171/JNS-07/07/0001. PMID 17639865
- [Background] Manninen PH, Balki M, Lukitto K, Bernstein M. Patient satisfaction with awake craniotomy for tumor surgery: a comparison of remifentanil and fentanyl in conjunction with propofol. Anesth Analg. 2006 Jan;102(1):237-42. doi: 10.1213/01.ANE.0000181287.86811.5C. PMID 16368836
- [Background] Whittle IR, Midgley S, Georges H, Pringle AM, Taylor R. Patient perceptions of "awake" brain tumour surgery. Acta Neurochir (Wien). 2005 Mar;147(3):275-7; discussion 277. doi: 10.1007/s00701-004-0445-7. PMID 15627921
- [Background] Khu KJ, Doglietto F, Radovanovic I, Taleb F, Mendelsohn D, Zadeh G, Bernstein M. Patients' perceptions of awake and outpatient craniotomy for brain tumor: a qualitative study. J Neurosurg. 2010 May;112(5):1056-60. doi: 10.3171/2009.6.JNS09716. PMID 19612973
- [Background] Manninen PH, Tan TK. Postoperative nausea and vomiting after craniotomy for tumor surgery: a comparison between awake craniotomy and general anesthesia. J Clin Anesth. 2002 Jun;14(4):279-83. doi: 10.1016/s0952-8180(02)00354-9. PMID 12088812
- [Background] Leslie K, Troedel S, Irwin K, Pearce F, Ugoni A, Gillies R, Pemberton E, Dharmage S. Quality of recovery from anesthesia in neurosurgical patients. Anesthesiology. 2003 Nov;99(5):1158-65. doi: 10.1097/00000542-200311000-00024. PMID 14576554
- [Background] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940
- [Background] Perks A, Chakravarti S, Manninen P. Preoperative anxiety in neurosurgical patients. J Neurosurg Anesthesiol. 2009 Apr;21(2):127-30. doi: 10.1097/ANA.0b013e31819a6ca3. PMID 19295391